CLINICAL TRIAL: NCT00182117
Title: Pilot Bleeding Study
Brief Title: Pilot Bleeding Study: Risk and Protective Factors Associated With Bleeding in the Hemodialysis Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Organization: McMaster University (Other)
Other Study IDs: Division of Nephrology Funds
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2006-01-24 (Estimated); Status verified 2005-09

CONDITIONS: Bleeding; End Stage Renal Disease
Keywords: bleeding; end stage renal disease; antiplatelet therapy; anticoagulant therapy; hemodialysis
MeSH Terms: conditions — Hemorrhage; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
This study is examining the risk and protective factors associated with bleeding in the hemodialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing hemodialysis

Exclusion Criteria:

* This is an observational study. No exclusion criteria required.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 490
Dates: Start 2003-10; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Rabbat, MD, Principal Investigator — Assistant Professor, Medicine
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada